CLINICAL TRIAL: NCT02436434
Title: The Effect of Intra-articular Pulsed Radiofrequency in Osteoarthritis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The effect is poor
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician, Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TriServiceGH
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Osteoarthritis
Keywords: Pulsed radiofrequency, osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pulsed radiofrequency (Active Comparator): Intra-articular pulsed radiofrequency (Neurotherm NT1000, Neurotherm Inc., USA) in treated joint
  Interventions: Device: pulsed radiofrequency (Neurotherm NT1000, Neurotherm Inc., USA)
- Sham pulsed radiofrequency (Sham Comparator): Sham intra-articular pulsed radiofrequency (Neurotherm NT1000, Neurotherm Inc., USA) in controlled joint
  Interventions: Device: pulsed radiofrequency (Neurotherm NT1000, Neurotherm Inc., USA)

INTERVENTIONS:
Device: pulsed radiofrequency (Neurotherm NT1000, Neurotherm Inc., USA) — Intra-articular pulsed radiofrequency (Neurotherm NT1000, Neurotherm Inc., USA) in treated joint

SUMMARY:
Pulsed radiofrequency (PRF) is designed to alleviate pain by delivering an electrical field and heat bursts at a temperature less than 42°C to neural tissue. In contrast with conventional radiofrequency, PRF is controlled below 42°C without damage to nerves and many studies have shown its benefits in pain relief for certain kinds of chronic pain conditions. For lessening pain of certain joint arthropathy, the direct nerve block by application of PRF is difficult and complicated because the supplying nerve of joint is complex or small. Hence, some authors perform intra-articular PRF on the chronic painful joint for example, knee osteoarthritis, atlantoaxial joint, cervical facet joint sacroiliac joint, scapholunate and shoulder joint and the excellent long-term effects are reported.

The purpose of this study is to investigate the effect of intra-articular PRF in osteoarthritis.

DETAILED DESCRIPTION:
Pulsed radiofrequency (PRF) is designed to alleviate pain by delivering an electrical field and heat bursts at a temperature less than 42°C to neural tissue. In contrast with conventional radiofrequency, PRF is controlled below 42°C without damage to nerves and many studies have shown its benefits in pain relief for certain kinds of chronic pain conditions. For lessening pain of certain joint arthropathy, the direct nerve block by application of PRF is difficult and complicated because the supplying nerve of joint is complex or small. Hence, some authors perform intra-articular PRF on the chronic painful joint for example, knee osteoarthritis, atlantoaxial joint, cervical facet joint sacroiliac joint, scapholunate and shoulder joint and the excellent long-term effects are reported.

However, the definite effect of intra-articular PRF for osteoarthritis from current published studies are insufficiently proved because of small patient numbers and lack of placebo-controlled design. The purpose of this study is to investigate the effect of intra-articular PRF in osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30-75 year-old
* Clear consciousness
* No receive steroid injection, hyaluronic acid, platelet rich plasma in past 6 months
* The pain (VAS) more than 4
* Symptom duration at least 6 months

Exclusion Criteria:

* Cancer
* Joint contracture
* Coagulopathy
* Pregnancy
* Status of Pacemaker
* Inflammation status
* Operative history of treated joint

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on1st, 2th, 4th, 8th,12th and 16th weeks after treatment. | Pre-treatment, 1st, 2th, 4th, 8th,12th and 16th weeks after treatment.
  Using the Visual analog scale (VAS) to measure the pain scale before treatment and multiple time frame after treatment.

SECONDARY OUTCOMES:
Change from baseline in severity of symptoms and functional status on1st, 2th, 4th, 8th,12th and 16th weeks after treatment. | Pre-treatment, 1st, 2th, 4th, 8th,12th and 16th weeks after treatment.
  Use the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) to measure the symptoms and functional status before treatment and multiple time frame after treatment.
Change from baseline of range of motion on1st, 2th, 4th, 8th,12th and 16th weeks after treatment. | Pre-treatment, 1st, 2th, 4th, 8th,12th and 16th weeks after treatment.
  Use the goniometer to measure the ROM before treatment and multiple time frame after treatment.
Change from baseline of strength on 4th, 8th,12th and 16th weeks after treatment. | Pre-treatment 4th, 8th,12th and 16th weeks after treatment.
  Use the isokinetic machine to measure the ROM before treatment and multiple time frame after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (2):
- Taiwan (2):
  - Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District
  - Tri-Service General Hospital, National Defense Medical Center,, Taipei, Neihu District

REFERENCES:
- [Background] Sluijter ME, Teixeira A, Serra V, Balogh S, Schianchi P. Intra-articular application of pulsed radiofrequency for arthrogenic pain--report of six cases. Pain Pract. 2008 Jan-Feb;8(1):57-61. doi: 10.1111/j.1533-2500.2007.00172.x. No abstract available. PMID 18211593
- [Background] Rahimzadeh P, Imani F, Faiz SH, Entezary SR, Nasiri AA, Ziaeefard M. Investigation the efficacy of intra-articular prolotherapy with erythropoietin and dextrose and intra-articular pulsed radiofrequency on pain level reduction and range of motion improvement in primary osteoarthritis of knee. J Res Med Sci. 2014 Aug;19(8):696-702. PMID 25422652
- [Background] Masala S, Fiori R, Raguso M, Morini M, Calabria E, Simonetti G. Pulse-dose radiofrequency for knee osteoartrithis. Cardiovasc Intervent Radiol. 2014 Apr;37(2):482-7. doi: 10.1007/s00270-013-0694-z. Epub 2013 Aug 14. PMID 23942592
- [Background] Karaman H, Tufek A, Kavak GO, Yildirim ZB, Uysal E, Celik F, Kaya S. Intra-articularly applied pulsed radiofrequency can reduce chronic knee pain in patients with osteoarthritis. J Chin Med Assoc. 2011 Aug;74(8):336-40. doi: 10.1016/j.jcma.2011.06.004. Epub 2011 Jul 23. PMID 21872812